### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | | Reporting and Analysis Plan (RAP) |

Title

: Reporting and Analysis Plan for 204706:

A single centre, single dose, open-label, randomized, 2-part, 2-way crossover study to determine the bioequivalence of levocetirizine oral disintegrating tablet given with water and without water compared to levocetirizine immediate release tablet in healthy Japanese male subjects

Compound Number

: GSK2074687 (Levocetirizine)

Effective Date

: 15-MAY-2018

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Pharmacology Study Report for Protocol 204706.
- This RAP is intended to describe the safety and pharmacokinetics analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

### RAP Author(s):

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Study statistician (Manager, Biostatistics Group 1, Biomedical Data Sciences Department, Japan) | | |
| PPD | | |
| Pharmacokineticist (Staff, Clinical Pharmacology Office, Japan) | 14-MAY-2018 | eSignature |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| CIL and OSL (Manager, Clinical Pharmacology Office, Medicines Development, Japan | 14-MAY-2018 | eSignature |
| PPD | | |
| DQL (Staff, Data Practice Group, Biomedical Data Sciences Department, Japan) | 15-MAY-2018 | eSignature |
| PPD | | |
| Clinical programmer (Manager, Statistical<br>Programming & Reporting Group, Biomedical<br>Data Sciences Department, Japan) | 15-MAY-2018 | eSignature |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Statistics Line approver (Associate Manager, Biostatistics Group 1, Biomedical Data Sciences Department, Japan) | 14-MAY-2018 | eSignature |
| Clinical Programming Line approver (Department Manager, Biomedical Data Sciences Department, Japan) | 14-MAY-2018 | eSignature |

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRODU | JCTION | | 6 |
| 2. | SUMMAR | Y OF KEY PRO | TOCOL INFORMATION | 6 |
| | 2.1. Ch | nanges to the Pro | otocol Defined Statistical Analysis Plan | 6 |
| | | | and Endpoint(s) | |
| | 2.4. St | atistical Hypothes | ses / Statistical Analyses | 8 |
| 3. | PLANNE | O ANALYSES | | 9 |
| | 3.1. Int | erim Analyses | | 9 |
| 4. | ANALYSI | S POPULATION | S | 9 |
| | | | ) | |
| 5. | | | DATA ANALYSES AND DATA HANDLING | |
| | | | Sub-group Display Descriptors | |
| | | | 3 | 10 |
| | 5.3. Ot | her Consideratio | ns for Data Analyses and Data Handling | |
| | Co | onventions | | 11 |
| 6. | STUDY P | OPULATION AN | ALYSES | 11 |
| - | | | | |
| 7. | SAFETY | ANALYSES | | 11 |
| | 7.1. Ac | lverse Events An | alyses | 11 |
| | 7.2. Cli | inical Laboratory | Analyses | 11 |
| | 7.3. Ot | her Safety Analy | ses | 12 |
| 8. | | COKINETIC AND | ALYSES | 12 |
| Ο. | | | kinetic Analyses | |
| | | | / Variables | |
| | 0. | 8.1.1.1. | | |
| | | • | Drug Concentration Measures Derived Pharmacokinetic Parameters | |
| | 0. | | | |
| | | , | Measure | |
| | | | n of Interest | |
| | | | for Intercurrent (Post-Randomization) Events | |
| | 8. | | Analyses / Methods | 13 |
| | | 8.1.5.1. | Statistical Methodology Specification | 13 |
| | | • | cokinetic Analyses | |
| | 8.2 | • | / Variables | |
| | | 8.2.1.1. | Drug Concentration Measures | |
| | | 8.2.1.2. | Derived Pharmacokinetic Parameters | |
| | | | Measure | |
| | _ | | n of Interest | |
| | | | for Intercurrent (Post-Randomization) Events | |
| | 8.2 | | Analyses / Methods | |
| | | 8251 | Statistical Methodology Specification | 16 |

| 9. | EXPLO | ORATOR) | Y ANALYSE | S | 16 |
|---|---|---|---|---|---|
| 10. | REFER | RENCES. | | | 17 |
| 11 | APPEN | NDICES | | | 18 |
| | 11.1. | | | I Deviation Management | |
| | 11.2. | | | le of Activities | |
| | 11.2. | 11 2 1 | Protocol D | efined Schedule of Events | 10 |
| | 11.3. | | | ment Windows | |
| | 11.4. | Appendix | x 4: Study P | hases and Treatment Emergent Adverse | |
| | | 11.4.1. | | ses | |
| | | 11.4.2. | | Emergent Flag for Adverse Events | |
| | 11.5. | | | splay Standards & Handling Conventions | |
| | | 11.5.1. | | Process | |
| | | 11.5.2. | | Standards | |
| | | 11.5.3. | | Standards for Pharmacokinetic | |
| | 11.6. | | | and Transformed Data | |
| | | 11.6.1. | General | | 23 |
| | | 11.6.2. | | ulation | |
| | | 11.6.3. | | | |
| | | 11.6.4. | Pharmacol | kinetic | 24 |
| | | 11.6.5. | Exploratory | / | 24 |
| | 11.7. | Appendix | | ng Standards for Missing Data | |
| | | 11.7.1. | Premature | Withdrawals | 25 |
| | | 11.7.2. | Handling o | f Missing Data | 25 |
| | | | 11.7.2.1. | Handling of Missing and Partial Dates | 25 |
| | | | 11.7.2.2. | Handling of Missing for Statistical Analysis of | |
| | | | | BE | 26 |
| | 11.8. | Appendix | x 8: Values | of Potential Clinical Importance | 27 |
| | | 11.8.1. | | Values | |
| | | 11.8.2. | ECG | | 28 |
| | | 11.8.3. | Vital Signs | | 28 |
| | 11.9. | | | ations & Trade Marks | |
| | | 11.9.1. | | ons | |
| | | 11.9.2. | | S | |
| | 11.10. | | | Data Displays | |
| | | | | ay Numbering | |
| | | | | nple Shell Referencing | |
| | | | | 2S | |
| | | | | Study Population Tables | |
| | | | | Safety Tables | |
| | | | | Pharmacokinetic Tables | |
| | | | | Pharmacokinetic Figures | |
| | | | | Exploratory Tables | |
| | | | | ICH Listings | |
| | | | | Non-ICH Listings | |
| | | 11 10 5 | | Non-ion Listings | |
| | | 11.10.3. | | Study Population Tables | |
| | | | | Safety Tables | |
| | | | 1 1. IU.D.J. | Pharmacokinetic Tables | 40 |

## 2018N384106\_00 204706

### CONFIDENTIAL

| 11.10.5.4. | Pharmacokinetic Figures | 47 |
|------------|------------------------------------|----|
| | Exploratory Tables | |
| | ICH Listings | |
| | Non-ICH Listings | |
| | ple Mock Shells for Data Displays. | |
| | p | • |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Pharmacology Study Report for Protocol.

| Revision Chronology | | |
|---------------------|-------------|----------|
| Version 00 | 15-MAY-2018 | Original |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 20/Apr/2018).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the bioequivalence between levocetirizine ODT (Orally Disintegrating Tablet) 5 mg (Test product) and levocetirizine IRT (Immediate Release Tablet) 5 mg (Reference product) in healthy Japanese male subjects | Plasma PK parameters of levocetirizine: AUC(0-t) and Cmax |
| Secondary Objectives | Secondary Endpoints |
| To assess the safety and tolerability following a single dose of levocetirizine 5 mg when given as levocetirizine ODT and levocetirizine IRT in healthy Japanese male subjects. | <ul> <li>Adverse events (AEs), changes from baseline in clinical laboratory tests, vital signs (blood pressure, pulse rate and body temperature), and 12-lead electrocardiogram (ECG).</li> <li>Plasma PK parameters of levocetirizine: AUC(0-inf), tmax, t1/2, %AUCex, CL/F, Vz/F, kel and MRT.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To assess the palatability questionnaire | The palatability questionnaire |

## 2.3. Study Design

## Overview of Study Design and Key Features

## Part 1 (Dosing of levocetirizine ODT with water)

- Single dose of levocetirizine ODT 5 mg x 1 with 150 mL of water in the fasted state
- Single dose of levocetirizine IRT 5 mg x 1 with 150 mL of water in the fasted state

| Group | n | Period 1 | Period 2 |
|-------|----|-------------------------|-------------------------|
| Α | 12 | Levocetirizine IRT 5 mg | Levocetirizine ODT 5 mg |
| | | (with water) | (with water) |
| В | 12 | Levocetirizine ODT 5 mg | Levocetirizine IRT 5 mg |
| | | (with water) | (with water) |

## Part 2 (Dosing of levocetirizine ODT without water)

- Single dose of levocetirizine ODT 5 mg x 1 without water in the fasted state
- Single dose of levocetirizine IRT 5 mg x 1 with 150 mL of water in the fasted state

| Group | n | Period 1 | Period 2 |
|-------|----|-------------------------|-------------------------|
| С | 12 | Levocetirizine IRT 5 mg | Levocetirizine ODT 5 mg |
| | | (with water) | (without water) |
| D | 12 | Levocetirizine ODT 5 mg | Levocetirizine IRT 5 mg |
| | | (without water) | (with water) |

| Design<br>Features | <ul> <li>This is a single centre, open-label, single dose, randomized, 2-way crossover study in healthy Japanese male subjects.</li> <li>This study consists of two parts: Part 1 compares dosing of levocetirizine ODT and levocetirizine IRT taken with 150 mL water in the fasted state, Part 2 compares dosing of levocetirizine ODT without water and levocetirizine IRT with 150 mL water in the fasted state.</li> <li>If subjects prematurely discontinue the study, additional replacement subjects may be recruited and assigned to the same treatment sequence at the discretion of the Sponsor in consultation with the investigator.</li> <li>If bioequivalence cannot be demonstrated in Part 1 and/or Part 2 because of an insufficient number of subjects, an add-on subject study will be performed using 12 (6 subjects in each group) or more subjects in each part.</li> </ul> |
|---|---|
| Dosing | All subjects will receive a single dose of levocetirizine 5 mg after an overnight fast (at least 10 hours) during the intervention period |
| Time & Events | Refer to Appendix 2: Schedule of Activities. |
| Treatment<br>Assignment | <ul> <li>In both parts (Part 1 and Part 2), total number of 24 subjects will be equally divided into two groups (12 subjects in each group) and will be randomized in a 1:1 ratio to one of two groups in each part.</li> <li>Subjects will participate either in Part 1 or Part 2 without overlapping.</li> </ul> |
| Interim<br>Analysis | No formal interim analyses are planned. |

## 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to test the bioequivalence of levocetirizine ODT 5 mg (with water or without water) relative to levocetirizine IRT 5 mg.

The null hypothesis is that the true ratio of the geometric mean of the levocetirizine ODT 5mg ( $\mu_{test}$ ) to the geometric mean of the levocetirizine IRT 5mg ( $\mu_{ref}$ ),  $\mu_{test}/\mu_{ref}$ , for each primary PK endpoint (AUC(0-t) and Cmax of levocetirizine), is either less than or equal to 0.80 or greater than or equal to 1.25. The alternative hypothesis is that the true ratio of the test treatment geometric mean to the reference treatment geometric mean is greater than 0.80 and less than 1.25.

Symbolically, this is expressed as follows:

 $H_0$ :  $\mu_{\text{test}}/\mu_{\text{ref}} \le 0.80$  or  $\mu_{\text{test}}/\mu_{\text{ref}} \ge 1.25$ ,

i.e., treatments are not bioequivalent.

Versus

 $H_1$ : 0.80 <  $\mu_{\text{test}}/\mu_{\text{ref}}$  < 1.25,

i.e., treatments are bioequivalent.

These hypotheses will be considered for levocetirizine ODT 5 mg with water or without water separately, relative to levocetirizine IRT 5 mg.

For each PK parameter designated as a primary endpoint (AUC(0-t) and Cmax), a two one-sided t-test (TOST) procedure [Schuirmann, 1987] with  $\alpha$ =0.05 for each one-sided test will be used to test this set of hypotheses. This is equivalent to requiring that a 90% interval for the true ratio of levocetirizine ODT 5 mg to levocetirizine IRT 5 mg geometric means ( $\mu_{test}/\mu_{ref}$ ) falls entirely within the range of 0.80 to 1.25. A judgment by 90% CI will be conducted in this study.

If the bioequivalence will not be shown above, ODT 5 mg will be accepted as bioequivalent where the point estimate for true ratio of levocetirizine ODT 5 mg to levocetirizine IRT 5 mg geometric mean ( $\mu_{test}/\mu_{ref}$ ) of AUC(0-t) and Cmax are within 0.90 - 1.11, according to the criteria described in the Japanese Guideline for Bioequivalence Studies of Generic Products (Japanese BE guideline) [Pharmaceutical and Food Safety Bureau, Evaluation and Licensing Division, Ministry of Health, Labour, 2012].

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal interim analyses are planned.

## 3.2. Final Analyses

The final analyses will be performed after the completion of the following sequential steps in each part respectively:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. Randomization codes have been distributed according to RandAll NG procedures.

As for an add-on subject study, the same sequential step above will be conducted.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Consisting of all participants screened in the study. | Study Population |
| Screening Failure | <ul> <li>Participants who sign the ICF in the study but are never<br/>subsequently randomized. All participants who sign the<br/>ICF have the screening test in the study.</li> </ul> | Study Population |
| Safety | <ul> <li>All randomized participants who take at least one dose of study treatment.</li> <li>Participants will be analyzed according to the treatment they actually received.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>Palatability</li><li>Questionnaire</li></ul> |
| Pharmacokinetic | <ul> <li>This population is defined as all participants administered at least one dose of study treatment and who have blood for plasma drug concentration sample taken and analyzed.</li> <li>Participants will be analyzed according to the treatment they actually received.</li> </ul> | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| Α | Levocetirizine ODT 5 mg | Levocetirizine ODT 5 mg | 1 |
| Α | Levocetirizine IRT 5 mg | Levocetirizine IRT 5 mg | 2 |
| В | Levocetirizine IRT 5 mg | Levocetirizine IRT 5 mg | 2 |
| В | Levocetirizine ODT 5 mg | Levocetirizine ODT 5 mg | 1 |

Randomized group (sequence) will be displayed as A or B for Part 1, and C (= A in RandAll NG) or D (= B in RandAll NG) for Part 2 according to the protocol.

### 5.2. Baseline Definitions

Baseline to be used in analysis is pre-dose in each period. For all endpoints, the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits

| Parameter | Study Asses | Baseline Used in | |
|---|---|---|---|
| | Screening | Data Display | |
| Safety | | | |
| Clinical Laboratory<br>Test (Hematology,<br>Clinical chemistry, and<br>Urinalysis) | Х | X | Day 1 (Pre Dose) |
| 12 Lead ECG & Vital<br>Signs | Х | Х | Day 1 (Pre Dose) |

Data of height, weight and BMI for demographic characteristics will be from screening visit.

Unless otherwise stated, if baseline data is missing, no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Reporting Standards for Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |

### 6. STUDY POPULATION ANALYSES

Study population analyses including analyses of subject's disposition, protocol deviations, demographic characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

### 8. PHARMACOKINETIC ANALYSES

The PK analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 8.1. Primary Pharmacokinetic Analyses

### 8.1.1. Endpoint / Variables

## 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Standards for Pharmacokinetic)

### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (version 6.3 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC (0-t)<br>(hr*ng/mL) | Area under the concentration-time curve from time zero time (pre-dose) to the time of last quantifiable concentration (AUC(0-t)) will be calculated by the linear trapezoidal method (i.e., Linear Trapezoidal Linear Interpolation calculation method in Phoenix WinNonlin). |
| Cmax<br>(ng/mL) | Maximum observed concentration will be obtained directly from the concentration-time data. |

### 8.1.2. Summary Measure

PK parameters of AUC(0-t) and Cmax are summary measures.

### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the PK population, unless otherwise specified.

### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

This section is not applicable, however, where a missing data for PK parameters will occur in a subject on period 1 or period 2, the subject data will be analyzed using the mixed effect model to evaluate the bioequivalence of PK parameter.

## 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

### **Endpoint / Variables**

AUC(0-t) and Cmax

### Model Specification

- Evaluation of BE will be performed for each part (Part 1 and Part 2) according to the criteria described in the Japanese BE Guideline.
- After log<sub>e</sub>-transformation, primary PK parameter(s) of levocetirizine given as levocetirizine ODT 5 mg or when given as levocetirizine IRT 5 mg will be analyzed using a mixed effects model fitting terms for treatment and period as fixed effects, also subjects as a random effect.
- The Kenward & Roger (KR) degrees of freedom approach will be used.
- Point estimates for the adjusted means on the log<sub>e</sub> scale, the mean difference between treatments and associated 90% confidence interval for the contrast (test-reference) will be constructed using the residual variance.
- The point estimate and confidence interval will then be exponentially back-transformed to obtain adjusted (least square) geometric means for each treatment, and point estimates and associated 90% confidence interval for the ratio test/reference.
- Two treatment are considered to be bioequivalent, if the 90% confidence intervals of the geometric mean ratio (μ<sub>test</sub>/μ<sub>ref</sub>) of AUC(0-t) and Cmax are within the acceptable range of 0.80 – 1.25.
- Estimates of within-subject variability (%CVw) for AUC (0-t) and Cmax of levocetirizine will also be provided.
- The within-subject coefficients of variation (%CVw) for AUC(0-t) and Cmax will be calculated based on the loge-normal distribution where:

%CVw= SQRT(exp(MSE)-1) \* 100

MSE is the residual mean squared error from the model

- If the bioequivalence will not be shown above, ODT 5 mg will be accepted as bioequivalent to IRT 5mg where the following condition is satisfied.
  - Point estimate for geometric mean ratio ( $\mu_{\text{test}}/\mu_{\text{ref}}$ ) of AUC(0-t) and Cmax are within 0.90 1.11.

### Add-on subject study

### **Endpoint / Variables**

- When an add-on subject study will be conducted, the data of two studies in each part would be combined for analysis.
- ODT 5 mg will be accepted as bioequivalent if the following condition is satisfied under the total pooled sample size of the main and add-on subject according to the criteria described in the Japanese BE Guideline.
  - $_{\odot}$  The 90% confidence intervals of the geometric mean ratio ( $\mu_{test}/\mu_{ref}$ ) of AUC(0-t) and Cmax are within the acceptable range of 0.80 1.25.
  - o If the bioequivalence will not be shown above, point estimate for geometric mean ratio  $(\mu_{test}/\mu_{ref})$  of AUC(0-t) and Cmax are within 0.90 1.11.
- After log<sub>e</sub>-transformation, primary PK parameter(s) of levocetirizine given as levocetirizine
  ODT 5 mg or when given as levocetirizine IRT 5 mg will be analyzed using a mixed effects
  model fitting terms for treatment, period and study (main or add-on subject study) as fixed
  effects, also subjects as a random effect.

## 8.2. Secondary Pharmacokinetic Analyses

## 8.2.1. Endpoint / Variables

### 8.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Standards for Pharmacokinetic)

### 8.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (version 6.3 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC (0-inf)<br>(hr*ng/mL) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC(0-inf)) will be calculated as follows: |
| | AUC(0-inf) = AUC(0-t) + C(t) / kel |
| %AUCex (%) | The percentage of AUC (0-inf) obtained by extrapolation (%AUCex) will be calculated as: |
| | %AUCex = [AUC(0-inf) - AUC(0-t)] / AUC(0-inf) x 100 |
| tmax (hr) | Time to first occurrence of Cmax will be obtained directly from the concentration-time data. |
| t1/2 (hr) | Apparent terminal phase half-life will be calculated as: |
| | t½ = In2 / kel |
| tlast (hr) | The time of the last measurable (positive) concentration. |
| kel<br>(lambda_z)<br>(1/hr) | The first order rate constant associated with the terminal (log-linear) portion of the curve. |
| lambda_z | The lower limit on time for values to be included in the calculation of kel. |

| Parameter | Parameter Description |
|---|---|
| lower (hr) | |
| lambda_z<br>upper (hr) | The upper limit on time for values to be included in the calculation of kel. |
| #pts | The number of time points used in computing kel. |
| R-square | Square of the correlation coefficient. |
| CL/F (L/hr) | Apparent clearance following oral dosing will be calculated as: |
| | CL/F = Dose / AUC (0-inf) |
| Vz/F (L) | Apparent volume of distribution following oral dosing will be calculated as: |
| | Vz/F = Dose / kel * AUC(0-inf) |
| MRT (hr) | Mean residence time will be calculated as follows: |
| | MRT = AUMC(0-inf) / AUC(0-inf) |

#### NOTES:

- Additional parameters may be included as required.
- kel is the terminal phase rate constant.
- C(t) is the last observed quantifiable concentration.
- AUMC is area under the moment curve.

## 8.2.2. Summary Measure

Derived PK parameters are shown in Section 8.2.1.2." Derived Pharmacokinetic Parameters" are summary measures.

## 8.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the PK population, unless otherwise specified.

### 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

This section is not applicable, however, where a missing data for PK parameters will occur in a subject on period 1 or period 2, the subject data will be analyzed using the mixed effect model to evaluate the bioequivalence of PK parameter.

## 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 8.2.5.1. Statistical Methodology Specification

### **Endpoint / Variables**

AUC(0-inf), tmax, kel, MRT

### **Model Specification**

- Same manner as Section 8.1.5.1. "Statistical Methodology Specification" for AUC(0-inf), kel, MRT.
- tmax will be analyzed with the non-parametric Wilcoxon Matched Pairs Method (Signed Rank Method) to compute point estimate and associated 90% confidence interval for the median difference, Levocetirizine ODT 5 mg – Levocetirizine IRT 5 mg, using normal approximation. Paired data of Levocetirizine ODT 5 mg and Levocetirizine IRT 5 mg will be used only and period effect will not be considered.

### Add-on subject study

- Same manner as Section 8.1.5.1. "Statistical Methodology Specification" for AUC(0-inf), kel, MRT.
- tmax will be analyzed with the non-parametric Wilcoxon Matched Pairs Method (Signed Rank Method) to compute point estimate and associated 90% confidence interval for the median difference, Levocetirizine ODT 5 mg – Levocetirizine IRT 5 mg, using normal approximation. Paired data of Levocetirizine ODT 5 mg and Levocetirizine IRT 5 mg will be used only and period effect and study effect (main or add-on subject study) will not be considered.

## 9. EXPLORATORY ANALYSES

The analysis of the palatability questionnaire will be based on the Safety population. The data will be summarized using descriptive statistics. All categorical responses will be summarized with counts and percentages. All ordinal data, e.g. ratings, will be summarized with mean, median, standard deviation, minimum, and maximum as well as counts and percentages of each rating. Palatability questionnaire data will also be listed.

## 10. REFERENCES

GlaxoSmithKline Document Numbers 2018N360906\_00 Study Protocol of 204678. A single centre, single dose, 2 part, open-label, randomized, 2-way crossover study to determine the bioequivalence of levocetirizine oral disintegrating tablet given with water and without water compared to levocetirizine immediate release tablet in healthy Japanese male subjects (Effective date: 20-Apr-2018)

Pharmaceutical and Food Safety Bureau, Evaluation and Licensing Division, Ministry of Health, Labour, and Welfare. Guideline for Bioequivalence Studies of Generic Products. Notification 0229 No.10. Feb-2012.

Schuirmann DJ. 1987. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. *J Pharmacokinet and Biopharm*, 15, 657-680.

# 11. APPENDICES

# 11.1. Appendix 1: Protocol Deviation Management

Details will be referred latest Protocol Deviation Management Plan and data handling will be decided prior to final data base release.

# 11.2. Appendix 2: Schedule of Activities

### 11.2.1. Protocol Defined Schedule of Events

| | | | Part 1 and Part 2 Intervention period (Period 1 and Period 2) | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>2</sup> | | | | | | | | Day 1 | | | | | | | Da | y 2 | Day 3 | Follow- |
| | | | Day -1 | Pre<br>dose | 0 h | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 9 h | 12 h | 16 h | 24 h | 36 h | 48 h |
| Informed consent | Х | | | | | | | | | | | | | | | | | | |
| Admission to unit | | X | | | | | | | | | | | | | | | | | |
| Height, Weight, Body<br>mass index (BMI) | х | | | | | | | | | | | | | | | | | | |
| Physical examination | Х | Х | X | | | | Х | | | | | | | | | Х | | Х | X |
| Serology test | Х | | | | | | | | | | | | | | | | | | |
| Clinical laboratory test1 | Х | | X | | | | | | | | | | | | | | | X | X |
| Urine drug screen | Х | | | | | | | | | | | | | | | | | | |
| 12-lead ECG | Х | | Х | | | | Х | | | | | | | | | | | Х | X |
| Vital signs | Х | | X | | | | X | | | | | | | | | Х | | Х | X |
| PK blood sampling | | | X | | X | Х | Х | X | Х | Х | X | X | X | Х | X | Х | Х | X | |
| Study intervention | | | | Х | | | | | | | | | | | | | | | |
| Palatability<br>Questionnaire <sup>4</sup> | | | | | | | | | | | | | | | | | | | |
| Adverse events | | | | <b>←</b> | | | | | | | | | | | | | | | <del></del> |
| Discharge from unit | | | | | | | | | | | | | | | | | | X | |

- 1. Clinical laboratory test: haematology, clinical chemistry, and urinalysis
- 2. Screening: up to 30 days prior to Day 1 of Period 1
- 3. Follow-up: 5-7 days post dose of Period 2
- 4. Palatability questionnaire will be administered to each subject within 10 minutes following dosing of ODT treatments only

## 11.3. Appendix 3: Assessment Windows

Not applicable

# 11.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

### 11.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to dosing by period.

| Study Phase | Definition |
|---------------|--------------------------------------------------------|
| Pre-Treatment | Date <= Day -1 in Period 1 |
| On-Treatment | Period 1: From Day 1 of Period 1 to Day 3 in Period 1. |
| | Period 2: From Day 1 of Period 2 to Day 3 in Period 2. |
| Follow-Up | After Day 3 in Period 2. |

### 11.4.2. Treatment Emergent Flag for Adverse Events

Adverse events will be classified according to the time of occurrence relative to start and/or stop date of the study treatment by period.

| Flag (Treatment State) | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date and Time in Period 1 |
| On treatment (Period 1) | <ul> <li>Dosing Start Date and Time in Period 1 ≤ AE Start Date and Time &lt; Study<br/>Treatment Start Date and Time in Period 2</li> </ul> |
| On treatment (Period 2) | Dosing Start Date and Time in Period 2 ≤ AE Start Date and Time < Follow-Up |
| Onset Time Since<br>First Dose | AE Onset Date and Time – Dosing Start Date and Time (if Dosing Start Date and Time > AE Onset Date and Time) |
| (Minute) | <ul> <li>AE Onset Date and Time - Dosing Start Date and Time +1 (if dosing Start Date<br/>and Time ≤ AE Onset Date and Time)</li> </ul> |
| | Missing otherwise |
| Onset Time Since<br>Last Dose<br>(Minute) | AE Start Date and Time – Most Recent Treatment Start Date and Time + 1 |
| Duration (Minute) | AE Resolution Date and Time – AE Onset Date and Time + 1 |

### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.
- If AE onset time is missing, the duration will be calculated in days.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

### 11.5.1. Reporting Process

| Software | |
|---|---|
| The currently supplementary | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : N/A |
| HARP Compound | HARP Compound : N/A |
| Analysis Datasets | Analysis Datasets |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated. | |

## 11.5.2. Reporting Standards

### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 11.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Office will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | No PK parameters derived by programmer are planned. |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters in GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. tmax will not be log <sub>e</sub> -transformed for summary statistics. |

## 11.6. Appendix 6: Derived and Transformed Data

### 11.6.1. General

### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < (Dosing Start Date) → Study Day = Ref Date (Dosing Start Date)</li>
- Ref Data ≥ (Dosing Start Date) → Study Day = Ref Date (Dosing Start Date) + 1

### 11.6.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - o Any subject with a missing day will have this imputed as day '15'.
  - o Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Reference date for age calculation will be from dosing start day.
- Reference date for calculation of age at screening will be from informed consent date.
- Analysis age group will be categorized (Years):
  - <=18, 19-64, 65-74, >=75
- Age will be categorized for EudraCT:

Adults (18-64 years)

## 11.6.3. Safety

#### **Adverse Events**

### **AE'S OF Special Interest**

N/A

### **Laboratory Assessments**

### Haematology

Platelet Count, RBC Count, Haemoglobin, Hematocrit, RBC Indices (MCV, MCH, MCH, %Reticulocytes), WBC count with Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils)

### **Clinical Chemistry**

BUN, Creatinine, Glucose (fasting), Potassium, Sodium, Calcium, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline phosphatise, Total and direct bilirubin, Total Protein

### **Laboratory Assessments**

### **Routine Urinalysis**

- Specific gravity, pH (assessed by dipstick)
- Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen by dipstick

### ECG (12-lead ECG)

ECG findings, ECG values (Heart rate, PR interval, QRS duration, QT interval, and QTcF intervals)

### **Vital Signs**

Pulse rate (Heart rate), Blood pressure (Systolic, Diastolic), Temperature

### 11.6.4. Pharmacokinetic

### PK parameters

### **Primary parameters**

AUC(0-t), Cmax

### Secondary parameters

AUC(0-inf), tmax, t1/2, %AUCex, CL/F, Vz/F, kel, MRT (tlast, lambda\_z lower, lambda\_z upper, #pts, R-square will be listed only)

### NQ, NC and ND

- If one or more non-quantifiable (NQ) values occur in a profile before the first measurable concentration, they will be assigned a value of zero concentration. For linear plots, zero concentration value(s) before the first measurable concentration will be included in the plot. For log-linear plots, zero concentration value(s) before the first measurable concentration will be assigned a missing value.
- If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be set to missing in the derivation of pharmacokinetic parameters, statistical analysis, and the individual subject plots.
- If two or more NQ values occur in succession between measurable concentrations, the profile will be
  deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of
  individual subject plots, these NQs will be set to 0, and the subsequent measurable concentrations will
  be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent
  measurable concentrations will be set to missing.
- NQs which occur after the last measurable concentration will be omitted (set to missing) in the derivation of pharmacokinetic parameters and from the individual subject plots.
- Individual's PK parameters reported as 'NC' (Not Calculable) or 'ND' (Not Determined) will be included in listings but omitted (set to missing) from figures, summaries and statistical analyses.

## 11.6.5. Exploratory

### **Palatability Questionnaire**

- Q1: to describe the taste of the product in subject's own words briefly
- Q2: to rate the palatability (acceptability of taste)
- Q3: to check all the descriptors (Sweet, Sour/tart, Bitter, Fruity, Nutty, Chalky, Medicinal)
- Q4: to rate the mouth feel
- Q5: to circle the number that best describes (5 score: Sweetness, Sour/tartness, Bitter)

# 11.7. Appendix 7: Reporting Standards for Missing Data

## 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as a subject has completed all phases of the study including the last follow-up visit as described in the protocol.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> </ul> |
| | Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.7.2.2. Handling of Missing for Statistical Analysis of BE

| Element | Reporting Detail |
|---|---|
| Imputation | <ul> <li>No imputation will be performed for missing data.</li> <li>Where a missing data for PK parameters (except for tmax) will occur in a subject on period 1 or period 2, the subject data will be analyzed using the mixed effect model to evaluate the bioequivalence of PK parameter</li> </ul> |

# 11.8. Appendix 8: Values of Potential Clinical Importance

# 11.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | n/I | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

Note: ↓ indicates a negative direction of the change from baseline.

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | µmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

Note: † indicates a positive direction of the change from baseline.

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 11.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc (QTcF) Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc (QTcF) | msec | | > 60 |

# 11.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate (Pulse Rate) | bpm | < 40 | > 110 |

# 11.9. Appendix 9: Abbreviations & Trade Marks

# 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| AUC | Area under concentration-time curve |
| AUC(0-inf) | Area under the concentration-time curve from time zero (pre-dose) extrapolated |
| ( | to infinite time |
| %AUCex | Percentage of AUC(0-inf) obtained by extrapolation |
| AUC(0-t) | Area under the concentration-time curve from pre-dose to last time of |
| , | quantifiable concentration within a subject across all treatments |
| BE | Bioequivalence |
| BMI | Body mass index |
| CI | Confidence Interval |
| CIL | Clinical Investigation Leader |
| CL/F | Apparent clearance following oral dosing |
| Cmax | Maximum observed concentration |
| CSR | Clinical Study Report |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DQL | Data Quality Leader |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| ICF | Informed Consent Form |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| LLQ | Lower Limit of Quantification |
| LS | Least Squar |
| MedDRA | Medical dictionary for regulatory activities |
| MSE | Mean Square Error |
| OSL | Operations and Science Leader |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| t1/2 | Terminal phase half-life |
| tmax | Time of occurrence of Cmax |
| TOST | Two one-sided t-test |

| Abbreviation | Description |
|--------------|-----------------------------------------------------------|
| Vz/F | Apparent volume of distribution after oral administration |

## 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

## 11.10. Appendix 10: List of Data Displays

## 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

Part 1:

| Section | Tables | Figures |
|------------------|--------------------|----------------|
| Study Population | 1.101 to 1.107 N/A | |
| Safety | 2.101 to 2.118 | N/A |
| Pharmacokinetic | 3.101 to 3.106 | 3.101 to 3.105 |
| Exploratory | 4.101 | N/A |
| Section | Listings | |
| ICH Listings | 101 to 138 | |
| Other Listings | 139 | |

Part 2:

| Section | Tables | Figures |
|------------------|----------------|----------------|
| Study Population | 1.201 to 1.207 | N/A |
| Safety | 2.201 to 2.218 | N/A |
| Pharmacokinetic | 3.201 to 3.206 | 3.201 to 3.205 |
| Exploratory | 4.201 | N/A |
| Section | Listi | Listings |
| ICH Listings | 201 to | 201 to 238 |
| Other Listings | 23 | 239 |

If an add-on subject study will be conducted, the data of two studies will be combined for analysis. The following numbering will be applied for RAP generated displays:

Part 1:

| Section | Tables | Figures |
|------------------|----------------|----------------|
| Study Population | 1.301 to 1.307 | N/A |
| Safety | 2.301 to 2.318 | N/A |
| Pharmacokinetic | 3.301 to 3.306 | 3.301 to 3.305 |
| Explanatory | 4.301 | N/A |
| Section | Listings | |
| ICH Listings | 301 to 338 | |
| Other Listings | 339 | |

## Part 2:

| Section | Tables | Figures |
|------------------|----------------|----------------|
| Study Population | 1.401 to 1.407 | N/A |
| Safety | 2.401 to 2.418 | N/A |
| Pharmacokinetic | 3.401 to 3.406 | 3.401 to 3.405 |
| Explanatory | 4.401 | N/A |

| Section | Listings |
|----------------|------------|
| ICH Listings | 401 to 438 |
| Other Listings | 439 |

## 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Exploratory | EXP_Fn | EXP_Tn | EXP_Ln |

### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 11.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| TR [X] | Topline Report |
| SAC [X] | Final Statistical Analysis Complete |

### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 11.10.4. Part 1

# 11.10.4.1. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.101 | Safety | CP_ES1 | Summary of Subject Disposition (Part 1) | Completed or withdrawn and the reason for withdrawal. | SAC [1] |
| 1.102 | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure (Part 1) | The number (%) of Randomized or screening failure subjects as the screening status, and the reason for screening failure. | SAC [1] |
| Protoc | ol Deviation | | | | |
| 1.103 | Safety | DV1 | Summary of Important Protocol Deviations (Part 1) | Data is from DV dataset. | SAC [1] |
| Study | Populations | | | | |
| 1.104 | Safety | SP1 | Summary of Study Populations (Part 1) | | SAC [1] |
| Demog | Demographics | | | | |
| 1.105 | Safety | DM3 | Summary of Demographic Characteristics (Part 1) | | TR [2] |
| 1.106 | Screened | DM11 | Summary of Age Ranges (Part 1) | Adults (18-64 years) | SAC [1] |
| 1.107 | Safety | DM5 | Summary of Race and Racial Combinations (Part 1) | | SAC [1] |

204706

## 11.10.4.2. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.101 | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 1) | | TR [2] |
| 2.102 | Safety | AE5A | Summary of All Adverse Events by System Organ Class and Maximum Intensity (Part 1) | | SAC [1] |
| 2.103 | Safety | AE1CP | Summary of All Drug-Related Adverse Events by<br>System Organ Class and Preferred Term (Part 1) | | SAC [1] |
| 2.104 | Safety | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity (Part 1) | | SAC [1] |
| 2.105 | Safety | AE1CP | Summary of Serious Adverse Events by System Organ Class (Part 1) | | SAC [1] |
| Labs | | | | | |
| 2.106 | Safety | LB1 | Summary of Chemistry Results (Part 1) | | SAC [1] |
| 2.107 | Safety | LB1 | Summary of Chemistry Changes from Baseline (Part 1) | | SAC [1] |
| 2.108 | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range (Part 1) | Worst Case Post-Baseline is not needed | SAC [1] |
| 2.109 | Safety | LB1 | Summary of Hematology Results (Part 1) | | SAC [1] |

204706

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.110 | Safety | LB1 | Summary of Hematology Changes from Baseline (Part 1) | | SAC [1] |
| 2.111 | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range (Part 1) | Worst Case Post-Baseline is not needed | SAC [1] |
| 2.112 | Safety | UR3b | Summary of Urinalysis (Glucose, Protein, Blood, Ketones) Data (Part 1) | | SAC [1] |
| 2.113 | Safety | LB1 | Summary of Urinalysis (Gravity and pH) (Part 1) | | SAC [1] |
| ECGs | | | | | |
| 2.114 | Safety | EG1 | Summary of ECG Findings (Part 1) | | SAC [1] |
| 2.115 | Safety | EG2 | Summary of ECG Values (Part 1). | | SAC [1] |
| 2.116 | Safety | EG2 | Summary of Change from Baseline in ECG Values (Part 1). | | SAC [1] |
| Vital Si | Vital Signs | | | | |
| 2.117 | Safety | VS1 | Summary of Vital Signs (Part 1) | | SAC [1] |
| 2.118 | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 1). | | SAC [1] |

## 11.10.4.3. Pharmacokinetic Tables

| Pharmacokinetic Tal |
|---------------------|

204706

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| PK Concentration Data | | | | | |
| 3.101 | PK | PK01: PKCT1 | Summary of Levocetirizine Plasma Concentration (ng/mL) (Part 1) | Summary statistics: N, n, Number of imputed, mean, 95% confidence interval, standard deviation, median, minimum, maximum | SAC [1] |
| Derive | PK Paramete | ers | | | |
| 3.102 | PK | PK03: PKPT1 | Summary of Levocetirizine Plasma Pharmacokinetic Parameters (non-transformed) (Part 1) | Summary statistics: N, n, Number of imputed, mean, 95% confidence interval, standard deviation, median, minimum, maximum | TR [2] |
| 3.103 | PK | PK05: PKPT3 | Summary of Levocetirizine Plasma Pharmacokinetic Parameters (loge-transformed) (Part 1) | Summary statistics: N, n, Number of imputed, geometric mean, 95% confidence interval for the geometric mean, standard deviation of logarithmically transformed data (SD(logs)), coefficient of variation (%CVb). | TR [2] |
| | | | | tmax is not included in this table. | |
| 3.104 | PK | Study Specific<br>(PK_T1) | Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (AUC(0-t) and Cmax) (Part 1) | PK Parameters: AUC(0-t), Cmax | TR [2] |
| 3.105 | PK | Study Specific<br>(PK_T1) | Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (AUC(0-inf), kel, MRT) (Part 1) | PK Parameters: AUC(0-inf), kel, MRT | TR [2] |
| 3.106 | PK | Study Specific (PK_T2) | Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (tmax) (Part 1) | PK Parameter: tmax. Non-parametric Wilcoxon Matched Pairs Method for median difference. | TR [2] |
# 11.10.4.4. Pharmacokinetic Figures

| Pharma | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentra | tion Plots | | | |
| 3.101 | PK | PK16b:<br>PKCF1x | Individual Levocetirizine Plasma Concentration-Time Plots by Subject (Linear and Semi-Log) (Part 1) | Paginate by Subject. Include line for LLQ along with footnote defining LLQ value (2.0 ng/mL) | SAC [1] |
| 3.102 | PK | PK16b:<br>PKCF1x | Individual Levocetirizine Plasma Concentration-Time<br>Plots by Treatment (Linear and Semi-Log) (Part 1) | Paginate by Treatment. Include line for LLQ along with footnote defining LLQ value (2.0 ng/mL) | SAC [1] |
| Mean / | Median Conce | entration Plots | | | |
| 3.103 | PK | PK17: PKCF2 | Mean (+SD) Levocetirizine Plasma Concentration-<br>Time Plots (Part 1) | Include the + SD bars at each time point. X-axis displays planned relative time Include line for LLQ along with footnote defining LLQ value (2.0 ng/mL) | TR [2] |
| 3.104 | PK | PK18: PKCF3 | Median Levocetirizine Plasma Concentration-Time Plots (Part 1) | | TR [2] |
| PK par | PK parameter Plots (Bioequivalence Analysis) | | | | |
| 3.105 | PK | Study Specific<br>(PK_F1) | Plot of Levocetirizine Treatment Ratio and 90%<br>CI for Bioequivalence Analysis on PK<br>Parameters (AUC(0-t) and Cmax) (Part 1) | PK Parameters: AUC(0-t), Cmax. Plot the comparison on the Y-axis and Ratio on X axis. | TR [1] |

## 11.10.4.5. Exploratory Tables

| Palatak | Palatability Questionnaire Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Palatab | ility Question | naire Tables | | | |
| 4.101 | Safety | Study Specific<br>(EXP_T1) | Summary of Palatability Questionnaire (Part 1) | Q2 to Q5. Summary statistics and frequency count will be performed for all questions except for Q3 of frequency only. | SAC [1] |

## 11.10.4.6. ICH Listings

Note: 'Inv.' in the standard displays will be replaced to 'Centre'.

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | misation | | | | |
| 101 | Safety | CP_TA2 | Listing of Randomised and Actual Treatments (Part 1) | | SAC [1] |
| Subjec | t Disposition | | | | |
| 102 | Safety | CP_ES10x | Listing of Reasons for Premature Withdrawal (Part 1) | | SAC [1] |
| 103 | Screening<br>Failure | ES7 | Listing of Reasons for Screening Failure (Part 1) | | SAC [1] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 104 | Safety | DV2 | Listing of Subjects with Important Protocol Deviations (Part 1) | | SAC [1] |
| 105 | Screened | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Part 1) | | SAC [1] |
| 106 | Safety | Study Specific<br>(SAFE_L1) | Listing of Subjects Excluded from PK Population (Part 1) | | SAC [1] |
| Demog | raphics | | | | |
| 107 | Safety | DM4 | Listing of Demographic Characteristics (Part 1) | Informed consent date is included. | SAC [1] |
| 108 | Screening<br>Failure | DM2 | Listing of Demographic Characteristics for Screening Failure Subjects (Part 1) | Informed consent date is included. | SAC [1] |
| 109 | Safety | DM10 | Listing of Race (Part 1) | | SAC [1] |
| 110 | Screening<br>Failure | DM10 | Listing of Race for Screening Failure Subjects (Part 1) | | SAC [1] |
| Medica | I Conditions | | | | |
| 111 | Screened | MH3 | Listing of Medical Conditions (Part 1) | | SAC [1] |
| Conco | mitant Medica | tions | | | |
| 112 | Screened | CP_CM4 | Listing of Concomitant Medications (Part 1) | | SAC [1] |
| 113 | Safety | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text (Part 1) | | SAC [1] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | ıre | | | | |
| 114 | Safety | EX4 | Listing of Exposure (Part 1) | | SAC [1] |
| Advers | e Events | | | | |
| 115 | Safety | CP_AE9 | Listing of All Adverse Event (Part 1) | | TR [2] |
| 116 | Safety | CP_AE9 | Listing of Serious Adverse Events (Part 1) | | TR [2] |
| 117 | Screening<br>Failure | CP_AE9 | Listing of Serious Adverse Events for Screening Failure Subject (Part 1) | | SAC [1] |
| 118 | Safety | CP_AE9 | Listing of Adverse Events Leading to Discontinuation of Investigational Product or Withdrawal from Study (Part 1) | | SAC [1] |
| 119 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 1) | | SAC [1] |
| 120 | Screened | AE2 | Listing of Relationship between System Organ Class, Preferred Term and Verbatim Text (Part 1) | | SAC [1] |
| LABS | | | | | |
| 121 | Safety | CP_LB6 | Listing of All Chemistry Data (Part 1) | Change from baseline is included. | SAC [1] |
| 122 | Safety | CP_LB6 | Listing of All Chemistry Data for Subjects with Potential Clinical Importance (Part 1) | | SAC [1] |
| 123 | Safety | CP_LB6 | Listing of All Hematology Data (Part 1) | Change from baseline is included. | SAC [1] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 124 | Safety | CP_LB6 | Listing of All Hematology Data for Subjects with Potential Clinical Importance (Part 1) | | SAC [1] |
| 125 | Safety | CP_LB6 | Listing of Urinalysis (Gravity and pH) Data (Part 1) | | SAC [1] |
| 126 | Safety | UR2b | Listing of Urinalysis (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen and microscopic examination) Data (Part 1) | | SAC [1] |
| Vital Si | gns | | | | |
| 127 | Safety | CP_VS5 | Listing of All Vital Signs (Part 1) | | SAC [1] |
| 128 | Safety | CP_VS5 | Listing of Change from Baseline in Vital Signs (Part 1) | | SAC [1] |
| 129 | Safety | CP_VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance (Part 1) | | SAC [1] |
| ECG | | | | | |
| 130 | Safety | CP_EG6 | Listing of ECG Findings (Part 1) | | SAC [1] |
| 131 | Safety | CP_EG4 | Listing of All ECG Values (Part 1) | | SAC [1] |
| 132 | Safety | CP_EG4 | Listing of Change from Baseline in ECG Values (Part 1) | | SAC [1] |
| 133 | Safety | CP_EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance (Part 1) | | SAC [1] |

204706

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Liver e | vent | | | | |
| 134 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting (Part 1) | | SAC [1] |
| 135 | Safety | MH3 | Listing of Medical Conditions for Subjects with Liver<br>Stopping Events (Part 1) | | SAC [1] |
| 136 | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part 1) | | SAC [1] |
| Pharma | acokinetics | | | | |
| 137 | PK | PK08: PKCL1x | Listing of Levocetirizine Plasma Concentration (Part 1) | | SAC [1] |
| 138 | PK | PK14: PKPL1x | Listing of Levocetirizine Plasma Pharmacokinetic Parameters (Part 1) | | SAC [1] |

## 11.10.4.7. Non-ICH Listings

| Non-IC | Non-ICH Listings | | | |
|---|---|---|---|---|
| No. Population IDSL / TST ID / Example Shell Title Programming Notes Deliveration Programming Notes Programming No | | | | |
| Palatak | ility Question | naire | | |
| 139 | Safety | Study Specific (EXP_L1) | Listing of Palatability Questionnaire (Part 1) | SAC [1] |

## 11.10.5. Part 2

# 11.10.5.1. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.201 | Safety | CP_ES1 | Summary of Subject Disposition (Part 2) | Completed or withdrawn and the reason for withdrawal. | SAC [1] |
| 1.202 | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure (Part 2) | The number (%) of Randomized or screening failure subjects as the screening status, and the reason for screening failure. | SAC [1] |
| Protoc | ol Deviation | | | | |
| 1.203 | Safety | DV1 | Summary of Important Protocol Deviations (Part 2) | Data is from DV dataset. | SAC [1] |
| Study I | Populations | | | | |
| 1.204 | Safety | SP1 | Summary of Study Populations (Part 2) | | SAC [1] |
| Demog | raphics | | | | |
| 1.205 | Safety | DM3 | Summary of Demographic Characteristics (Part 2) | | TR [1] |
| 1.206 | Screened | DM11 | Summary of Age Ranges (Part 2) | Adults (18-64 years) | SAC [1] |
| 1.207 | Safety | DM5 | Summary of Race and Racial Combinations (Part 2) | | SAC [1] |

204706

## 11.10.5.2. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.201 | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 2) | | TR [1] |
| 2.202 | Safety | AE5A | Summary of All Adverse Events by System Organ Class and Maximum Intensity (Part 2) | | SAC [1] |
| 2.203 | Safety | AE1CP | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Part 2) | | SAC [1] |
| 2.204 | Safety | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity (Part 2) | | SAC [1] |
| 2.205 | Safety | AE1CP | Summary of Serious Adverse Events by System Organ Class (Part 2) | | SAC [1] |
| Labs | | | | | |
| 2.206 | Safety | LB1 | Summary of Chemistry Results (Part 2) | | SAC [1] |
| 2.207 | Safety | LB1 | Summary of Chemistry Changes from Baseline (Part 2) | | SAC [1] |
| 2.208 | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range (Part 2) | Worst Case Post-Baseline is not needed | SAC [1] |
| 2.209 | Safety | LB1 | Summary of Hematology Results (Part 2) | | SAC [1] |

204706

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.210 | Safety | LB1 | Summary of Hematology Changes from Baseline (Part 2) | | SAC [1] |
| 2.211 | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range (Part 2) | Worst Case Post-Baseline is not needed | SAC [1] |
| 2.212 | Safety | UR3b | Summary of Urinalysis (Glucose, Protein, Blood, Ketones) Data (Part 2) | | SAC [1] |
| 2.213 | Safety | LB1 | Summary of Urinalysis (Gravity and pH) (Part 2) | | SAC [1] |
| ECGs | | | | | |
| 2.214 | Safety | EG1 | Summary of ECG Findings (Part 2) | | SAC [1] |
| 2.215 | Safety | EG2 | Summary of ECG Values (Part 2). | | SAC [1] |
| 2.216 | Safety | EG2 | Summary of Change from Baseline in ECG Values (Part 2). | | SAC [1] |
| Vital Si | gns | | | | |
| 2.217 | Safety | VS1 | Summary of Vital Signs (Part 2) | | SAC [1] |
| 2.218 | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 2). | | SAC [1] |

## 11.10.5.3. Pharmacokinetic Tables

## **Pharmacokinetic Tables**

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| PK Cor | K Concentration Data | | | | |
| 3.201 | PK | PK01: PKCT1 | Summary of Levocetirizine Plasma Concentration (ng/mL) (Part 2) | Summary statistics: N, n, Number of imputed, mean, 95% confidence interval, standard deviation, median, minimum, maximum | SAC [1] |
| Derive | d PK Paramete | ers | | | |
| 3.202 | PK | PK03: PKPT1 | Summary of Levocetirizine Plasma Pharmacokinetic Parameters (non-transformed) (Part 2) | Summary statistics: N, n, Number of imputed, mean, 95% confidence interval, standard deviation, median, minimum, maximum | TR [1] |
| 3.203 | PK | PK05: PKPT3 | Summary of Levocetirizine Plasma Pharmacokinetic Parameters (loge-transformed) (Part 2) | Summary statistics: N, n, Number of imputed, geometric mean, 95% confidence interval for the geometric mean, standard deviation of logarithmically transformed data (SD(logs)), coefficient of variation (%CVb). | TR [1] |
| | | | | tmax is not included in this table. | |
| 3.204 | PK | Study Specific (PK_T1) | Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (AUC(0-t) and Cmax) (Part 2) | PK Parameters: AUC(0-t), Cmax | TR [1] |
| 3.205 | PK | Study Specific (PK_T1) | Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (AUC(0-inf), kel, MRT) (Part 2) | PK Parameters: AUC(0-inf), kel, MRT | TR [1] |
| 3.206 | PK | Study Specific<br>(PK_T2) | Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (tmax) (Part 2) | PK Parameter: tmax. Non-parametric Wilcoxon Matched Pairs Method for median difference. | TR [1] |

## 11.10.5.4. Pharmacokinetic Figures

| Pharma | acokinetic Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentra | tion Plots | | | |
| 3.201 | PK | PK16b:<br>PKCF1x | Individual Levocetirizine Plasma Concentration-Time Plots by Subject (Linear and Semi-Log) (Part 2) | Paginate by Subject. Include line for LLQ along with footnote defining LLQ value (2.0 ng/mL) | SAC [1] |
| 3.202 | PK | PK16b:<br>PKCF1x | Individual Levocetirizine Plasma Concentration-Time Plots by Treatment (Linear and Semi-Log) (Part 2) | Paginate by Treatment. Include line for LLQ along with footnote defining LLQ value (2.0 ng/mL) | SAC [1] |
| Mean / | Median Conce | entration Plots | | | |
| 3.203 | PK | PK17: PKCF2 | Mean (+SD) Levocetirizine Plasma Concentration-<br>Time Plots (Part 2) | Include the + SD bars at each time point. X-axis displays planned relative time Include line for LLQ along with footnote defining LLQ value (2.0 ng/mL) | TR [1] |
| 3.204 | PK | PK18: PKCF3 | Median Levocetirizine Plasma Concentration-Time Plots (Part 2) | | TR [1] |
| PK par | ameter Plots ( | Bioequivalence A | nalysis) | | |
| 3.205 | PK | Study Specific<br>(PK_F1) | Plot of Levocetirizine Treatment Ratio and 90% CI for Bioequivalence Analysis on PK Parameters (AUC(0-t) and Cmax) (Part 2) | PK Parameters: AUC (0-t), Cmax. Plot the comparison on the Y-axis and Ratio on X axis. | TR [1] |

## 11.10.5.5. Exploratory Tables

| Palatab | Palatability Questionnaire Tables | | | | |
|---|---|---|---|---|---|
| No. | o. Population IDSL / TST ID / Example Shell Title Programming Notes | | | | Deliverable<br>[Priority] |
| Palatab | ility Question | naire Tables | | | |
| 3.206 | Safety | Study Specific<br>(EXP_T1) | Summary of Palatability Questionnaire (Part 2) | Q2 to Q5. Summary statistics and frequency count will be performed for all questions except for Q3 of frequency only. | SAC [1] |

## 11.10.5.6. ICH Listings

Note: 'Inv.' in the standard displays will be replaced to 'Centre'.

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | p. Population IDSL / TST ID / Example Shell Title | | | Programming Notes | Deliverable<br>[Priority] |
| Rando | misation | | | | |
| 201 | 01 Safety CP_TA2 Listing of Randomised and Actual Treatments (Part 2) | | | | SAC [1] |
| Subjec | t Disposition | | | | |
| 202 | Safety | CP_ES10x | Listing of Reasons for Premature Withdrawal (Part 2) | | SAC [1] |
| 203 | Screening<br>Failure | ES7 | Listing of Reasons for Screening Failure (Part 2) | | SAC [1] |

| ICH Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 204 | Safety | DV2 | Listing of Subjects with Important Protocol Deviations (Part 2) | | SAC [1] |
| 205 | Screened | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Part 2) | | SAC [1] |
| 206 | Safety | Study Specific<br>(SAFE_L1) | Listing of Subjects Excluded from PK Population (Part 2) | | SAC [1] |
| Demog | raphics | | | | |
| 207 | Safety | DM4 | Listing of Demographic Characteristics (Part 2) | Informed consent date is included. | SAC [1] |
| 208 | Screening<br>Failure | DM2 | Listing of Demographic Characteristics for Screening Failure Subjects (Part 2) | Informed consent date is included. | SAC [1] |
| 209 | Safety | DM10 | Listing of Race (Part 2) | | SAC [1] |
| 210 | Screening<br>Failure | DM10 | Listing of Race for Screening Failure Subjects (Part 2) | | SAC [1] |
| Medica | l Conditions | | | | |
| 211 | Screened | MH3 | Listing of Medical Conditions (Part 2) | | SAC [1] |
| Conco | mitant Medica | tions | | | |
| 212 | Screened | CP_CM4 | Listing of Concomitant Medications (Part 2) | | SAC [1] |
| 213 | Safety | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text (Part 2) | | SAC [1] |

| ICH Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposi | ure | | | | |
| 214 | Safety | EX4 | Listing of Exposure (Part 2) | | SAC [1] |
| Advers | e Events | | | | |
| 215 | Safety | CP_AE9 | Listing of All Adverse Event (Part 2) | | TR [1] |
| 216 | Safety | CP_AE9 | Listing of Serious Adverse Events (Part 2) | | TR [1] |
| 217 | Screening<br>Failure | CP_AE9 | Listing of Serious Adverse Events for Screening Failure Subject (Part 2) | | SAC [1] |
| 218 | Safety | CP_AE9 | Listing of Adverse Events Leading to Discontinuation of Investigational Product or Withdrawal from Study (Part 2) | | SAC [1] |
| 219 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 2) | | SAC [1] |
| 220 | Screened | AE2 | Listing of Relationship between System Organ Class, Preferred Term and Verbatim Text (Part 2) | | SAC [1] |
| LABS | | | | | |
| 221 | Safety | CP_LB6 | Listing of All Chemistry Data (Part 2) | Change from baseline is included. | SAC [1] |
| 222 | Safety | CP_LB6 | Listing of All Chemistry Data for Subjects with Potential Clinical Importance (Part 2) | | SAC [1] |
| 223 | Safety | CP_LB6 | Listing of All Hematology Data (Part 2) | Change from baseline is included. | SAC [1] |

| ICH Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 224 | Safety | CP_LB6 | Listing of All Hematology Data for Subjects with Potential Clinical Importance (Part 2) | | SAC [1] |
| 225 | Safety | CP_LB6 | Listing of Urinalysis (Gravity and pH) Data (Part 2) | | SAC [1] |
| 226 | Safety | UR2b | Listing of Urinalysis (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen and microscopic examination) Data (Part 2) | | SAC [1] |
| Vital Si | gns | | | | |
| 227 | Safety | CP_VS5 | Listing of All Vital Signs (Part 2) | | SAC [1] |
| 228 | Safety | CP_VS5 | Listing of Change from Baseline in Vital Signs (Part 2) | | SAC [1] |
| 229 | Safety | CP_VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance (Part 2) | | SAC [1] |
| ECG | | | | | |
| 230 | Safety | CP_EG6 | Listing of ECG Findings (Part 2) | | SAC [1] |
| 231 | Safety | CP_EG4 | Listing of All ECG Values (Part 2) | | SAC [1] |
| 232 | Safety | CP_EG4 | Listing of Change from Baseline in ECG Values (Part 2) | | SAC [1] |
| 233 | Safety | CP_EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [1] |

204706

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Liver e | vent | | | | |
| 234 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting (Part 2) | | SAC [1] |
| 235 | Safety | MH3 | Listing of Medical Conditions for Subjects with Liver<br>Stopping Events (Part 2) | | SAC [1] |
| 236 | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part 2) | | SAC [1] |
| Pharma | acokinetics | | | | |
| 237 | PK | PK08: PKCL1x | Listing of Levocetirizine Plasma Concentration (Part 2) | | SAC [1] |
| 238 | PK | PK14: PKPL1x | Listing of Levocetirizine Plasma Pharmacokinetic Parameters (Part 2) | | SAC [1] |

## 11.10.5.7. Non-ICH Listings

| Non-IC | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Programming Notes | Deliverable<br>[Priority] | |
| Palatab | Palatability Questionnaire | | | | |
| 239 | Safety | Study Specific (EXP_L1) | Listing of Palatability Questionnaire (Part 2) | | SAC [1] |

204706

# 11.11. Appendix 11: Example Mock Shells for Data Displays

Study specific mock shells are shown only.

204706

Example: Study Specific (PK\_T1) Page 1 of n

Protocol: 204706 Population: PK

Table X.XX

Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (AUC(0-t) and Cmax) (Part X)

| Parameter | N | Treatment | n | Geometric LS Mean | Ratio<br>[1] | 90% CI of the<br>Ratio | %CVw<br>[2] |
|---|---|---|---|---|---|---|---|
| AUC(0-t) (hr*ng/mL) | XX | Levocetirizine ODT 5 mg | XX | xxx.xx | xx.xx | (x.xxx, x.xxx) | XX.X |
| (III IIg/ IIII) | | Levocetirizine IRT 5 mg | xx | xxx.xx | | | |
| Cmax (ng/mL) | xx | Levocetirizine<br>ODT 5 mg | xx | xxxx.xx | xx.xx | (xx.xxx,<br>xx.xxx) | XX.X |
| | | Levocetirizine<br>IRT 5 mg | XX | xxxx.xx | | | |

<sup>[1]</sup> Ratio = Geometric LS Mean of Levocetirizine ODT 5 mg / Geometric LS Mean of Levocetirizine IRT 5 mg

<sup>[2] %</sup>CVw = sqrt[exp(MSE) - 1] \* 100

204706

Example: Study Specific (PK\_T2) Page 1 of n

Protocol: 204706 Population: PK

Table X.XX
Summary of Bioequivalence Analysis on Pharmacokinetic Parameters (tmax) (Part X)

| Parameter | N | Treatment | n | Median | n | Median<br>Difference | 90% CI of the<br>Difference |
|---|---|---|---|---|---|---|---|
| tmax (hr) | XX | Levocetirizine<br>ODT 5 mg | XX | xxxx.xx | XX | xx.xx | (xx.xxx,<br>xx.xxx) |
| | | Levocetirizine IRT 5 mg | XX | XXXX.XX | | | , |

Note: tmax will be analyzed with the non-parametric Wilcoxon Matched Pairs Method (Signed Rank Method) to compute point estimate and associated 90% confidence interval for the median difference, Levocetirizine ODT 5 mg - Levocetirizine IRT 5 mg, using normal approximation.


204706

Example: Study Specific (PK F1)

Protocol: 204706 Population: PK

Figure X.XX

Plot of Levocetirizine Treatment Ratio and 90% CI for Bioequivalence Analysis on PK Parameters (AUC(0-t) and Cmax) (Part X)



Ratio and 90% CI

Note: Ratio = Geometric LS Mean of Levocetirizine ODT 5 mg / Geometric LS Mean of Levocetirizine IRT 5 mg

AUC(0-t) (hr\*ng/mL), Cmax (ng/mL)


204706

Example: Study Specific (EXP T1)

Protocol: 204706
Population: Safety

Table X.XX
Summary of Palatability Questionnaire (Part X)

| Questions | | ODT 5mg<br>(N=XX) |
|--------------------------------|----------------------|-------------------|
| Q2. Palatability Rate | n<br>Mean | XX<br>x.x |
| | SD | X.XX |
| | Median | x.x |
| | Min. | Х |
| | Max. | X |
| | n | X |
| | 1 Unacceptable | x (xx%) |
| | 2 Neutral/Acceptable | x (xx%) |
| | 3 Very good | x (xx%) |
| Q3. All Description Associated | n | Х |
| | Bitter | x (xx%) |
| | Chalky | x (xx%) |
| | Fruity | x (xx%) |
| | Medicinal | x (xx%) |
| | Nutty | x (xx%) |
| | Sour | x (xx%) |
| | Sweet | x (xx%) |

Q4. Mouth Feel Rate, Q5a. Best Description (Sweetness), Q5b. Best Description (Sour/tartness), Q5c. Best Description (Bitter). Summary statistics and frequency count with % will be performed for all questions except for Q3.


204706

Example: Study Specific (EXP L1)

Protocol: 204706 Population: SP

Listing X.XX
Listing of Subjects Palatability Questionnaire (Part X)

| <pre>Treatment/ Site Id./</pre> | Age(y)/<br>Sex/ | Q1 | Q2 | Q3 | Q4 | Q5 | | |
|---|---|---|---|---|---|---|---|---|
| Unique Subject Id. | Race/<br>Assessor | | | | | a | b | С |
| Levocetirizine ODT 5mg/ | 26/<br>Male/<br>White/<br>Subject | xxx | 1:Unaccepta<br>ble | Sweet,<br>Fruity | 2:Neutral/Acc eptable | 1 | 1 | 3 |
| Levocetirizine IRT<br>5mg/<br>PPD | 39/<br>Male/<br>White/<br>Subject | xxx | 2:Neutral/A cceptable | Bitter | 3: Very good | 3 | 2 | 1 |

#### Note:

- Q1. Please briefly describe the taste of the product in your own words (one word, short phrase descriptions are acceptable)
- Q2. Please rate the palatability (acceptability of taste) of the product by checking a rating.
- Q3. Please check all the descriptors that apply to the product. (Multiple Answer allowed)
- Q4. Please rate the mouth feel of the product by checking a rating.
- Q5. Please circle the number that best describes your perception of each attribute: a=Sweetness b=Sour/tartness c=Bitter


204706

Example: Study Specific (SP L1)

Protocol: 204706
Population: Safety

Listing X.XX
Listing of Subjects Excluded from PK population (Part X)

Age(y)/

Treatment/

Site Id./ Sex/ PΚ Unique Subject Race Population Id. PPD 26/ Ν Male/ White 39/ Ν Male/ White